CLINICAL TRIAL: NCT00180427
Title: VERRARI - "Are Ventricular Arrhythmic Episodes Reduced by Rate Response in ICDs?"
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Guidant Corporation (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: Version vom 01.03.2001
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation

INTERVENTIONS:
Device: ICD

SUMMARY:
"The purpose of this study is to evaluate the influence of the rate response function of implantable cardioverter defibrillators (ICDs) on the frequency of ventricular arrhythmias in patients with an ICD."

DETAILED DESCRIPTION:
"Background: Studies have shown that bradycardia and irregular heart rates may increase the incidence of ventricular arrhythmias. Regularizing the heart rate and avoiding bradycardias by rate responsive pacing may be a way to reduce these arrhythmias.

This is a prospective, open-label, randomized multicenter study. Inclusion criteria: Patients with an indication for an ICD according to the AHA/ACC-guidelines who get a rate response system and have more than 5 % rate adaptive pacing during a one month screening phase may be included if they have given written informed consent. Rate adaptive pacing must not be contraindicated, patients must be able to perform a 6 min walk test, must not be NYHA IV and should have a life expectancy of more than 18 months.

Patients will be randomly assigned to 6 months of rate responsive pacing followed by 6 months of no rate responsive pacing, vice versa respectively. At 6 and 12 months follow ups, ICD stored data, arrhythmic episodes, medication, anamnesis, quality of life, 6 min walktest, echocardiographic parameters and optionally spiroergomatry will be evaluated and compared."

ELIGIBILITY:
Inclusion Criteria:

* indication for an ICD according to ACC/AHA guidelines
* ICD with rate response function implanted
* at least 5% rate response ventricular pacing during the one month screening phase
* signed informed patient consent"

Exclusion Criteria:

* rate responsive pacing contraindicated
* patient not able to perform 6 min walktest
* heart failure NYHA IV
* life expectancy below 18 months"

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75
Dates: Start 2001-06; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
frequency of ventricular arrhythmias at 6 and 12 months follow ups

SECONDARY OUTCOMES:
medication, anamnesis, quality of life, 6 min walktest, echocardiographic parameters and optionally spiroergomatry at 6 and 12 months follow ups,

CONTACTS AND LOCATIONS:
Overall Officials: Michael Niehaus, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Medizinische Klinik der Medizinischen Hochschule, Hanover, Germany